CLINICAL TRIAL: NCT06692036
Title: Adaptive Blood Purification for the Treatment of Patients With Septic Shock: a Multicenter, Open-label, Randomized, Parallel Controlled Study
Brief Title: Adaptive Blood Purification for the Treatment of Patients With Septic Shock
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Chao Yang Hospital (Other)
Collaborators: China-Japan Friendship Hospital (Other); Peking University First Hospital (Other); Beijing Hospital (Other Government); Air Force Military Medical University, China (Other); Beijing Jishuitan Hospital (Other); Chinese PLA General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Capital'sFunds2024-1-2031
Record Dates: First submitted 2024-10-22; First posted 2024-11-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2024-10

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (standard treatment) (No Intervention): Patients in the control group received standard treatment by the "Surviving sepsis campaign: international guidelines for management of sepsis and septic shock 2021".
- Intervention group (standard treatment + ABP) (Experimental): Intervention Type: Patients in the intervention group, based on standard treatment, received two 6-hour adaptive blood purification (ABP) treatments within 24 hours after enrollment, that is, patients did not indicate renal replacement therapy (RRT), only plasma filtration-adsorption (PFAD) therapy is used to adsorb inflammatory factors; for patients with acute kidney injury (AKI) and meeting RRT indications, PFAD-RRT treatment is used.
  Interventions: Other: Adaptive Blood Purification (ABP)

INTERVENTIONS:
Other: Adaptive Blood Purification (ABP) — Patients in the intervention group, based on standard treatment, received two 6-hour adaptive blood purification (ABP) treatments within 24 hours after enrollment, that is, patients did not indicate renal replacement therapy (RRT), only coupled plasma filtration-adsorption (PFAD) therapy is used to adsorb inflammatory factors; for patients with acute kidney injury (AKI) and meeting RRT indications, PFAD-RRT treatment is used.
  Arms: Intervention group (standard treatment + ABP)

SUMMARY:
There is a lack of evidence in the efficacy of extracorporeal blood purification (EBP) to reduce the mortality rate in septic shock. We have designed the EABPSS (Efficacy of Adaptive Blood Purification for Septic Shock) study to confirm whether adaptive blood purification (ABP) intervention could confer a clinical benefit. In this multicenter, open-label, randomized controlled trial, We are recruiting a total of 276 patients with septic shock. Eligible patients who provide informed consent will be randomly assigned in a 1:1 ratio to either the control group or the intervention group. Patients in the control group will receive standard care according to the Surviving Sepsis Guidelines. Patients in the intervention group will receive two 6-hour sessions of ABP treatment within 24 hours of enrollment, based on standard care. ABP is a novel, adaptive EBP strategy proposed by our research team, specifically, for patients with septic shock do not require renal replacement therapy (RRT), plasma filtration-adsorption (PFAD) will be used alone, and for patients with septic shock and acute kidney injury meeting RRT indications, a combination of PFAD-RRT will be employed. The primary endpoint of this study is all-cause mortality at 90 days after enrollment. Secondary endpoints of the study include the declining proportion of serum cytokines such as TNF-α, IL-4, IL-6, IL-8, IL-10, and HMGB1 within 24 hours after enrollment. Additionally, the study will evaluate the improvement of Sequential Organ Failure Assessment score on day 7 post-enrollment, as well as the 30-day mortality rate.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients admitted to intensive care unit (ICU), 18 years old ≤ age ≤ 82 years old;
2. Meeting the diagnostic criteria for septic shock (Sepsis 3.0), and the onset time of septic shock ≤ 24 hours;
3. Systemic inflammatory response syndrome (SIRS) ≥ 3 points;
4. Sequential organ failure assessment (SOFA) ≥ 6 points;
5. Voluntarily sign the informed consent form before the trial, and agree to participate in all visits, examinations, and treatments according to the requirements of the research plan.

Exclusion Criteria:

1. Patients who have received blood purification treatment within 1 week for any reason;
2. Patients with congenital or acquired immunodeficiency diseases, or those who have received organ transplantation;
3. Patients who have received immunosuppressive drugs (mycophenolate, cyclophosphamide, FK506, etc.) within 28 days before enrollment;
4. Patients who received continuous treatment (≥ 3 days) with more than 10 mg/day of prednisolone (or other hormones at equivalent doses) within 28 days before enrollment;
5. Patients with active bleeding (requiring blood transfusion > 3 units in the past 24 hours);
6. Patients with malignant tumors, those who cannot remove the lesions (such as surgical patients who cannot undergo surgical treatment);
7. End-stage organ failure (end-stage pulmonary heart disease, brain death, chronic liver disease combined with hepatic encephalopathy);
8. Platelet count < 30×10^9/L or neutrophil count < 0.5×10^9/L;
9. Patients who require supportive treatment due to acute pulmonary embolism or severe congestive heart failure;
10. The mean arterial blood pressure (MAP) cannot be maintained ≥ 65 mmHg after receiving vasoactive drugs and fluid resuscitation treatment;
11. Patients who have participated or participated in another clinical study within 28 days before enrollment;
12. Patients who are allergic to extracorporeal circulation materials, perfusion device materials or have a history of other severe allergies, or those who have heparin-associated thrombocytopenia;
13. Patients who are inappropriate for participating, such as pregnant or lactating women, patients with severe mental and neurological diseases, and those with a history of alcoholism that cannot be terminated.

Ages: 18 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality at day 90 | The follow-up time ends on the 90th day after patient enrollment.
  The primary endpoint is all-cause mortality at day 90 after enrollment.

SECONDARY OUTCOMES:
Declining proportion of serum cytokines | From enrollment to the end of first 24 hours.
  The declining proportion (DP %) of serum cytokines such as TNF-α, IL-4, IL-6, IL-8, IL-10, and HMGB1 within 24 hours after enrollment (DP % = (CytokineH0 - CytokineH24)/CytokineH0 ), H0 is the serum cytokine level measured at the time of enrollment; H24 is the serum cytokine level measured at 24h after enrollment).
Improvement of SOFA score | The follow-up time ends on the 7th day after patient enrollment.
  Improvement of sequential organ failure assessment score (SOFA) on the 7th day after enrollment.
All-cause mortality at day 30 | The follow-up time ends on the 30th day after patient enrollment.
  30-day all-cause mortality rate after enrollment.
Duration of stay | The follow-up time ends on the 90th day after patient enrollment.
  The duration of stay in the intensive care unit and in the hospital.
Mortality rate | The follow-up time ends on the 90th day after patient enrollment.
  The mortality rate within the intensive care unit and the hospital.
Requirement of RRT | The follow-up time ends on the 90th day after patient enrollment.
  The requirement of renal replacement therapy (RRT) at both day 30 and day 90 after enrollment.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Chao Yang Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
EABPSS (Efficacy of Adaptive Blood Purification for Septic Shock) study aims to confirm whether adaptive blood purification (ABP) intervention could confer a clinical benefit.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 2026.1.1-2028.12.31
Access Criteria: Researchers who focus on extracorporeal blood purification for the treatment of septic shock will be able to access the IPD and supporting information. And they will access the relevant data needed in the Case Report Form according to the visitor's research plan. By sending email to the research group, fill in the plan of the research scheme, and the feasibility of the scheme will be evaluated by the research group. If the evaluation is passed, the researcher will be granted access.

REFERENCES:
- [Derived] Jia H, Li X, Zheng Y, Cui N, Ronco C, Li W. Efficacy of Adaptive Blood Purification for Septic Shock (EABPSS): protocol for a randomised, multicentre, parallel controlled study. BMJ Open. 2025 Oct 20;15(10):e107311. doi: 10.1136/bmjopen-2025-107311. PMID 41120165